CLINICAL TRIAL: NCT03134053
Title: Assessment of the Effect of Extracorporeal Shock Waves on Hypertrophy Scar
Brief Title: Effect of Extracorporeal Shock Waves on Hypertrophy Scar
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mackay Memorial Hospital (Other)
Responsible Party: Principal Investigator, Li-Ru Chen,MD, MD, Mackay Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16MMHIS025e
Record Dates: First submitted 2017-04-19; First posted 2017-04-28 (Actual); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Hypertrophy; Scar
Keywords: hypertrophy scar; burn
MeSH Terms: conditions — Cicatrix, Hypertrophic; Burns | interventions — Extracorporeal Shockwave Therapy; Massage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- extracorporeal shock-wave (Experimental)
  Interventions: Device: extracorporeal shock-wave
- massage (Sham Comparator)
  Interventions: Other: massage

INTERVENTIONS:
Device: extracorporeal shock-wave — to treat painful and retracting scars
  Arms: extracorporeal shock-wave
Other: massage — to treat painful and retracting scars
  Arms: massage

SUMMARY:
Assess the effect of extracorporeal shock waves on hypertrophy scar

DETAILED DESCRIPTION:
Prolonged and abnormal scarring after trauma, burns and surgical procedures often results in functional and cosmetic deformities. A wide variety of treatments have been advocated for pathologic scars regression. Unfortunately, the reported efficacy has been variable.Unfocused extracorporeal shock wave therapy is a feasible and non-intensive treatment. And it is an emerging option for the treatment of painful and retracting scars.

Administration of ESWT appears to result in significant improvements in scar clinical appearance, mobility and subjective pain. Clinical data were mirrored by histologic changes in connective tissue appearance and scar vascularization. Extracorporeal shock wave therapy is also an effective and conservative treatment for patients with aesthetic and functional sequela from burn scars. It is a feasible, cost-effective, well-tolerated treatment that can be used in the management of post-burn pathologic scars after the patients are briefed on the practical aspects of the treatment procedure.

ELIGIBILITY:
Inclusion Criteria:

1. aged between 18 ~ 65 years old;
2. at least 4 weeks since onset of onset of wound;
3. healing wound with at least 6 scores in Modified Vancouver Scar Scale for more than four weeks
4. the most important of all, read and signed the inform concern of this study.

Exclusion Criteria:

1. patients with open wound;
2. oxygen dependent
3. having evidence of cognitive deficit;
4. having local infection, severe inflammation or otherwise lesion that is not suggestive for ESWT;
5. patient with serious medical problems, as uncontrolled hypertension, coagulopathy, recent severe hemorrhage, neoplasm, severe hepatic disease, epilepsy, cutaneous pathology, mental retardation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2017-10-01 (Estimated); Primary Completion 2017-12-01 (Estimated); Study Completion 2019-06-01 (Estimated)

PRIMARY OUTCOMES:
change from baseline thick of scar | immediately post intervention, 1 month after, and 3 months
  sonography for thick of scar

SECONDARY OUTCOMES:
change from baseline Modified Vancouver Scar Scale | immediately post intervention, 1 month after, and 3 months
  questionnaires of Modified Vancouver Scar Scale for scar measure
change from baseline Visual analogue scores (VAS) | immediately post intervention, 1 month after, and 3 months
  Visual analogue scores (VAS) for pain
change from baseline skin color | immediately post intervention, 1 month after, and 3 months
  DermaLab Combo series for skin color
change from baseline Patient Scar Assessment Scale (POSAS) | immediately post intervention, 1 month after, and 3 months
  questionnaires of Patient Scar Assessment Scale (POSAS) for scar measure

CONTACTS AND LOCATIONS:
Locations (1):
- Mackay Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No